CLINICAL TRIAL: NCT06435000
Title: An Observational Study in Subjects to Follow the Progression of Stargardt Disease Type 1 (STGD1) Caused by Bi-Allelic Autosomal Recessive Mutations in the ATP Binding Cassette Subfamily A Member 4 (ABCA4) Gene
Brief Title: An Observational Study in Subjects to Follow the Progression of Stargardt Disease Type 1 (STGD1) Caused by Bi-Allelic Autosomal Recessive Mutations in the ABCA4 Gene
Acronym: POLARIS
Status: Recruiting | Type: Observational
Sponsor: Splice Bio (Industry)
Responsible Party: Sponsor
Other Study IDs: SB-CS-001
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-08

CONDITIONS: Stargardt; Stargardt's Disease; Stargardt Disease; STGD1
Keywords: POLARIS; Splicebio; STGD1; ABCA4
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal saliva swab to determine a minimum of two pathogenic or likely pathogenic mutations in the ABCA4 gene to genetically confirm the disease, as per eligibility criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an Observational Study to Follow the Progression of Stargardt Disease Type 1 (STGD1) Caused by Bi-Allelic Autosomal Recessive Mutations in the ABCA4 Gene

This is a multicenter study which will enroll approximately 75 subjects

DETAILED DESCRIPTION:
Comprehensive knowledge of a disease is essential to the design and conduct of well-controlled, interventional clinical trials. Understanding of the disease state is important for identifying the patient population for a clinical trial, study duration, and selection of clinically meaningful endpoints.

Observational studies play an important role in the understanding of rare diseases and facilitating effective development of potential therapies. To support clinical research, observational studies can help define the clinical features of a rare disease, rate of progression, pathophysiology, and other important factors. Further, following the course of a disease over time allows investigators to identify demographic variables, genotypic and phenotypic features, and other characteristics that may correlate with disease and outcomes in the absence of treatment. Thus, observational studies are useful in guiding the design of therapeutic studies, including selection of the patient population, trial duration, and the types of outcome measures to evaluate efficacy and safety.

Results of a natural history study evaluating the progression of atrophy secondary to Stargardt Disease have been published using retrospective and prospective cohorts of patients (ProgStar, Strauss et al., 2016).

In summary, the current study is a prospective observational study of patients with STGD1, the aim of which is to further enhance understanding of disease progression and structural and functional markers that can be used to evaluate the efficacy and safety of therapeutic interventions, especially in light of advancements in imaging technology.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written consent
2. Are male or female aged 12-65 years old
3. Have a diagnosis of STGD1 caused by bi-allelic likely pathogenic or pathogenic variants in the ABCA4 gene confirmed genotypically by an accredited genotyping laboratory
4. Have a history of STGD1 progression within the last 2 years, in the opinion of the investigator.
5. Eligible eye(s) must have:

   1. BCVA of between 24-88 ETDRS letters, inclusive (20/20 - 20/320 Snellen equivalent, 0.0-1.2 logMAR) at the Screening Visit.
   2. Clinical evidence of a macular lesion phenotypically consistent with Stargardt Disease.
   3. Fundus autofluorescence (FAF) measurement of definitely decreased autofluorescence (DDAF) as measured by the Central Reading Center (CRC).
   4. Total lesion must be imaged in its entirety.
   5. All total lesion borders must be ≥300 microns from all image edges.
6. Eligible eye(s) must have clear ocular media and adequate pupillary dilation, including no allergy to dilating eyedrops, to permit good quality retinal imaging.

Exclusion Criteria:

1. Are an immediate family member (e.g., child, sibling) of the Sponsor or study site personnel.
2. Have any concurrent ocular disease that would affect study procedures or outcomes (e.g., cataracts; subjects can be enrolled 90 days after successful cataract surgery) in eligible eyes.
3. Have two likely pathogenic or pathogenic variants (not STGD1) in autosomal recessive inherited retinal dystrophy (IRD) genes or a single likely pathogenic or pathogenic variant in autosomal dominant or X-linked IRD genes.
4. Have had any intraocular surgery or thermal laser within 90 days of study entry or any prior thermal laser in the macular region within the eligible eye(s).
5. Have any major surgical procedure within 30 days of the Screening Visit or planned or anticipated major surgery during the study period.
6. Are unwilling to stop taking the following products at Screening and throughout the study:

   1. Supplements containing vitamin A or beta-carotene, liver-based products.
   2. Prescription oral retinoids.
7. Have actively participated in an investigational therapy study or have received any investigational therapy within 90 days of the Screening Visit or 5 half-lives, whichever is longer. Note: any ophthalmic history of gene therapy, stem cell therapy, surgical implantation of prosthetic retinal chips, or intravitreal or sub-retinal injections exclude the subject from study participation.
8. Have known serious allergies to the fluorescein dye that might be used to measure intraocular pressure (IOP), ocular dilating drops, topical ocular anesthetic, or any history of anaphylaxis reaction.
9. Have a history of amblyopia in the eligible eye(s).
10. Have any significant ocular or non-ocular disease/disorder (or medication and/or laboratory test abnormalities) which, in the opinion of the investigator and with concurrence of the Medical Monitor, may either put the subject at risk because of participation in the study, may influence the results of the study, or affect the subject's ability to participate in the study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected that have a genetic and clinical diagnosis of STGD1 and fulfil all other entry criteria.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Document disease progression based on change from baseline in lesion size as measured by DDAF on FAF imaging | 96 weeks

SECONDARY OUTCOMES:
Change from baseline in ellipsoid zone (EZ) area as measured by SD-OCT | 96 weeks
Change from baseline in BCVA using ETDRS | 96 weeks
Change from baseline in LLVA using ETDRS | 96 weeks
Change from baseline in retinal sensitivity based on macular microperimetry | 96 weeks
Change from baseline in contrast sensitivity scores | 96 weeks
Change from baseline using Patient Reported Outcome Questionnaires | 96 weeks

CONTACTS AND LOCATIONS:
Locations (20):
- United States (14):
  - Shiley Eye Institute, San Diego, California
  - UCHealth Sue Anschutz-Rodgers Eye Center, Aurora, Colorado
  - Vitreo Retinal Associates, Gainesville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Wilmer Eye Institute, Johns Hopkins University MD 21287, Baltimore, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Kellogg Clinical Research Center, Ann Arbor, Michigan
  - Columbia University Medical Center, New York, New York
  - CUIMC/Edward S. Harkness Eye Institute, New York, New York
  - Duke Eye Center, Durham, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
  - University of Wisconsin, Madison, Madison, Wisconsin
- Germany (2):
  - Universitätsklinikum Bonn, Klinik für Augenheilkunde, Bonn
  - University Eye Hospital Tübingen, Tübingen
- United Kingdom (4):
  - Moorfields Eye Hospital, London, London
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University of Manchester - The Old St Mary's Hospital, Manchester
  - Oxford Eye Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No
Sponsor will wait until data fully analyzed and published before considering sharing

REFERENCES:
- See also: SpliceBio — https://splice.bio/clinical/